CLINICAL TRIAL: NCT06308783
Title: Effects of Diaphragmatic Breathing and Global Postural Reeducation on Stress and Sleep Quality in Healthy University Students
Brief Title: Diaphragmatic Breathing and Global Postural Reeducation on Stress and Sleep Quality in University Students
Acronym: RPGBREATH23
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFranciscoVitoriaRPGBREATH23
Record Dates: First submitted 2024-02-05; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Stress; Sleep Disturbance
Keywords: diaphragmatic breathing; global posture reeducation; stress; sleep quality
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: One group receives Diaphragmatic Breathing, one group receives Global Postural Reeducation, and the other group receives no intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diaphragmatic Breathing (Experimental): Diaphragmatic breathing, also known as deep breathing, is based on breathing slowly and widely, expanding the abdomen and then the ribs on inspiration and emptying as much air as possible on exhalation.
  Interventions: Other: Diaphragmatic Breathing
- Global Postural Reeducation (Experimental): Global Postural Re-education (GPR) is a technique described by Philippe Souchard that is based on the active and sustained stretching of muscle chains by performing specific postures. Breathing plays a fundamental role in the development of exercise, influencing the structures of the body and its functioning.
  Interventions: Other: Global Postural Reeducation
- Control Group (No Intervention): No treatment

INTERVENTIONS:
Other: Diaphragmatic Breathing — 10 minutes each day during 6 weeks, before sleeping.
  Arms: Diaphragmatic Breathing
Other: Global Postural Reeducation — 10 minutes each day during 6 weeks, before sleeping.
  Other Names: GPR
  Arms: Global Postural Reeducation

SUMMARY:
Introduction: Nowadays, the reduction of perceived stress and the improvement of sleep quality are considered fundamental aspects in the quality of life of both healthy subjects and patients with disease. Stress has become a pandemic in recent years due to the socio-labor demands faced by society. On the other hand, it has a direct relationship with the quality of sleep, its influence being bidirectional. In this regard, several tools have been reported for the management of these conditions. These include strategies such as yoga, mindfulness, diaphragmatic breathing (DR) or Pilates. On the other hand, other proposals such as global postural reeducation (GPR) lack evidence in the management of these conditions.

Objectives: Compare the effects of a diaphragmatic breathing self-management program with global postural reeducation on stress and sleep quality in university students.

Method: The study will be carried out with physiotherapy students of the University Francisco de Vitoria. The participants will be randomly divided into three groups: GPR group, DR group and control group. Perceived stress (Perceived Stress Scale - PSS14) and reported sleep quality (Pittsburgh Sleep Quality Index - PSQI) will be measured three times throughout the study: pre-intervention, 3 weeks after the start of the intervention and post-intervention. The intervention will last 6 weeks, during which time all participants will be required to complete the 5 Grade Scale (5GS) each morning. The GPR group will perform; Frog to the ground posture, while the DR group will follow a set breathing protocol at a 4/6 rhythm. Both GPR and DR will be performed 10 minutes before going to sleep.

Ethical considerations:

The principles of the 1964 Declaration of Helsinki will be followed. The proposed interventions are non-invasive, based on the combination of mild physical activity tools, body awareness and relaxation techniques.

The dependent variables to be measured are based on clinimetric aspects, without any harm to the participants.

Subjects will be asked to participate on a voluntary basis and may withdraw from the study at any time.

DETAILED DESCRIPTION:
MATERIAL AND METHODS Type of study This work will be an analytical, experimental, longitudinal and prospective study, unblinded. The patients were randomly divided into 3 groups, one of which was a control group.

This study will be conducted in accordance with the 1964 Helsinki declaration.

Sample The target population of the study will be university students who suffer from stress. The accessible population will be physiotherapy students of the Francisco de Vitoria University.

Method of selection and assignment of participants to each group Before selecting our sample, we will divide the future participants into different groups with simple randomization.

To obtain the sample we will go through the physiotherapy classes of the UFV, explaining our project and providing each person with a QR code.

There will be a control group and two experimental groups (global posture reeducation and diaphragmatic breathing). The participants will not know which group they belong to until the day of the start of the intervention.

Variables

The independent variables of the study are:

* Global posture reeducation
* Diaphragmatic breathing

The dependent variables are:

* Stress
* Quality of sleep

Tools and measurements Stress The level of stress will be measured before and after the intervention using a validated questionnaire both in its original format and in its Spanish format.

Sleep quality To assess and measure the participants; sleep quality, we will use a questionnaire. The Pittsburgh Sleep Quality Index (PSQI) is the most commonly used tool in clinical and research to assess sleep quality. It proven valid, as well as its translation into Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over 18 years of age.
* Physiotherapy students of Francisco de Vitoria University.
* Ability to understand written and oral Spanish.
* Ability to communicate in Spanish or French.

Exclusion Criteria:

* < 18 years of age Cognitive disorders (psychiatric or mental).
* Problems when understanding instructions.
* Follow-up of a stress-focused treatment (medication, psychological therapy, meditation, etc.).
* Smokers.
* Pregnant women.
* Pathologies (rheumatic, neurological, cardiovascular, respiratory, visceral, tumor, fibromyalgia, physical handicap etc.).
* Serious accident or recent surgery.
* Sleep disorders (apnea...).
* Practice of a daily exercise similar to the intervention (Pilates, Yoga, tai chi, qi gong, etc.).
* Not undergoing any other intervention during the investigation.
* Suffering from stress lower than 29/56 on the PSS14 questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-07-18 (Estimated)

PRIMARY OUTCOMES:
Stress | First measure one day before starting the intervention, second measure 3 weeks after starting the intervention and third measure 6 weeks after starting the intervention (last day of intervention)
  Perceived Stress Scale Questionnaire
Sleep Quality | First measure one day before starting the intervention, second measure 3 weeks after starting the intervention and third measure 6 weeks after starting the intervention (last day of intervention)
  Pittsburgh Sleep Quality Index Questionnaire

SECONDARY OUTCOMES:
Sleep Quality | Up to 6 weeks.
  5 Grade Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Roldán Ruiz, PhD, Principal Investigator — Universidad Francisco de Vitoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hopper SI, Murray SL, Ferrara LR, Singleton JK. Effectiveness of diaphragmatic breathing for reducing physiological and psychological stress in adults: a quantitative systematic review. JBI Database System Rev Implement Rep. 2019 Sep;17(9):1855-1876. doi: 10.11124/JBISRIR-2017-003848. PMID 31436595
- [Result] Ferreira GE, Barreto RG, Robinson CC, Plentz RD, Silva MF. Global Postural Reeducation for patients with musculoskeletal conditions: a systematic review of randomized controlled trials. Braz J Phys Ther. 2016 Apr 1;20(3):194-205. doi: 10.1590/bjpt-rbf.2014.0153. PMID 27437710